CLINICAL TRIAL: NCT04319809
Title: Object Finder for a Retinal Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minnesota HealthSolutions (Industry)
Collaborators: Johns Hopkins University (Other); Second Sight Medical Products (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MHS-OF01
Record Dates: First submitted 2020-03-16; First posted 2020-03-24 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa; Argus II retinal prosthesis system
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: This is a small sample open label feasibility study for an object recognition and localization system based on machine learning
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Device feasibility (Experimental): To investigate the utility of a device adaptation allowing Argus II users to detect the presence and location of desired objects. Performance of the unaided Argus II system will be compared with performance using the system augmented with object recognition.
  Interventions: Device: Object recognition subsystem

INTERVENTIONS:
Device: Object recognition subsystem — The object recognition subsystem is an add-on to the Argus II retinal prosthesis system. in the early stage of the study the subsystem will run on a separate processor; in the later stage the subsystem will run in the Argus II user's video processing unit.

SUMMARY:
The proposed project seeks to provide object recognition as a feature in a retinal implant system. Participants will be able to direct an object recognition application to find a desired object in the field of view of the head-mounted camera, and to direct the participant's view towards it through the presentation of a recognizable icon. A prototype system will be developed and evaluated in human subjects in phase I. A full system implementation and a second phase of the trial will be completed in phase II.

DETAILED DESCRIPTION:
The investigators propose to add an object-finding feature to a retinal prosthesis system. To use this feature, the participant will enable a special mode and input the desired object from a set of pre-programmed object types. Imagery from the visible light camera in the system eyeglasses will be processed using object recognition software as the participant scans their head across the room scene. When the object is identified in the scene by the processor, a flashing icon will be output to the epiretinal array in the appropriate position to guide the participant to the physical location of the object. Once located, the system will track the location of the object.

There will be two phases to the human subjects evaluation, each run initially through simulations in sighted human subjects, followed by tests in Argus II participants. In phase 1, system evaluation in human subjects at Johns Hopkins UNiversity (JHU) will explore performance in representative tasks and compare prosthetic visual performance without and with the new object finding feature. An important aspect of the evaluation will be the comparison of different icons and presentation modes to assist participants in locating and reaching objects. In phase 2, the system will be integrated into the Argus II video processing unit (VPU), and JHU will conduct human trials that include functional testing of the integrated prototype in representative environments and optimizing the ergonomics of the system, e.g. simultaneous finding and tracking of multiple objects/icons.

ELIGIBILITY:
Inclusion Criteria:

* For healthy volunteers: Vision corrected to 20/25, good general health
* For retinitis pigmentosa (RP) patients: End-stage retinitis pigmentosa, recipient of an Argus II retinal prosthesis system

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gislin Dagnelie, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available from the investigative team, following initial publication of the results
Supporting Information: Study Protocol, SAP
Time Frame: Spring 2022 onward
Access Criteria: Any researchers wit ha legitimate reason for wishing to re-analyze the data or compare them to study data collected in similar experiments

RESULTS

PARTICIPANT FLOW:
Groups:
- Argus II Users: Blind individuals previously implanted with the Argus II retinal prosthesis system were invited to join the study. Data were collected in 4 participants ranging in age from 61 to 90 years old. One participant was female, all identified as white, non-hispanic.
- Legally Blind Individuals: Individuals with profound visual impairment (best corrected visual acuity worse than 20/500) were invited to join the study. Data were collected in 5 participants ranging in age from 31 to 54 years old. One participant was female, all identified as white, non-hispanic.
Period: Overall Study
Arm/Group | Argus II Users | Legally Blind Individuals
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: See enrollment group descriptions
Groups:
- Total: Total of all reporting groups
Arm/Group | Argus II Users | Legally Blind Individuals | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 6
  >=65 years | 3 | 0 | 3
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 77 [66 to 87] | 35 [32 to 50] | 54 [34 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 5 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Performance (Completion Time) Locating a Cell Phone and a Person
Description: This outcome measure compares time to task completion without and with modalities of the subsystem for both a stationary and mobility task. For the stationary task, participants were seated in front of a table and a cell phone was placed randomly at the center of one of ten rectangular zones. Participants were asked to find and put their hand on the location of the cell phone. The time of the response was recorded (and the distance from the cell phone, which is a separate primary outcome). For the mobility task, participants were asked to find a target person in an otherwise empty room with dark walls. Once the participant got within arm's length, the target person would initiate a handshake. The time and number of steps (a separate primary outcome) were recorded. If the person wasn't found within 5 minutes, the task was stopped and scored as incomplete.
Time Frame: Time in seconds to complete task. Stationary task time was time to placing hand on the table with the cell phone and mobility task time was time to handshake with the target person.
Population: Blind individuals previously implanted with the Argus II retinal prosthesis system were invited to join the study. Data were collected in 4 participants. Individuals with profound visual impairment (best corrected visual acuity worse than 20/500) were invited to join the study. Data were collected in 5 participants.
Measure: Mean (Standard Deviation); unit: time (s)
Groups:
- Argus II Users: To investigate the utility of a device adaptation allowing Argus II users to detect the presence and location of desired objects. Performance of the unaided Argus II system will be compared with performance using the system augmented with object recognition. Performance will be compared for Argus II Users and Legally Blind Individuals.
  Object recognition subsystem: The object recognition subsystem is an add-on to the Argus II retinal prosthesis system. in the early stage of the study the subsystem will run on a separate processor; in the later stage the subsystem will run in the Argus II user's video processing unit.
- Legally Blind Individuals: To investigate the utility of a device adaptation allowing Legally Blind Individuals to detect the presence and location of desired objects. Performance of the object finder system will be compared with performance using the system augmented with object recognition. Performance will be compared for Argus II Users and Legally Blind Individuals.
Arm/Group | Argus II Users | Legally Blind Individuals
Number analyzed (Participants) | 4 | 5
time (s)
  Stationary, Normal Camera | 47 (16.6) | 11 (13.5)
  Stationary, Icon | 30 (6.1) | 23 (9.7)
  Stationary, Tone | 26 (6.6) | 21 (10.4)
  Stationary, Speech | 19 (4.7) | 26 (18.1)
  Stationary, Normal Camera plus Tone | 24 (1.7) | 16 (17.3)
  Stationary, Normal Camera plus Speech | 27 (5.6) | 12 (9.4)
  Stationary, Tone plus Icon | 27 (2.9) | 22 (10.7)
  Stationary, Speech plus Icon | 27 (5.1) | 35 (33.1)
  Stationary, Tactile | 6 (2.0) | 6 (2.0)
  Mobility, Normal Camera | 135 (3.7) | 9 (15.6)
  Mobility, Icon | 37 (10.2) | 44 (86.1)
  Mobility, Tone | 35 (.9) | 17 (4.3)
  Mobility, Speech | 28 (6.6) | 15 (1.9)
  Mobility, Normal Camera plus Tone | 29 (9.1) | 6 (6.4)
  Mobility, Normal Camera plus Speech | 27 (11.4) | 9 (9.1)
  Tone plus Icon | 36 (1.6) | 8 (4.9)
  Speech plus Icon | 38 (10.5) | 12 (8.8)

2. Primary Outcome: Accuracy (Distance From Target)
Description: This outcome measure compares task completion (accuracy to a target) without and with modalities of the subsystem for both a stationary and mobility task. For the stationary task, participants were seated in front of a table and a cell phone was placed randomly at the center of one of ten rectangular zones. Participants were asked to find and put their hand on the location of the cell phone. The distance to the cell phone in centimeters was recorded. For the mobility task, participants were asked to find a target person in an otherwise empty room with dark walls. Once the participant got within arm's length, the target person would initiate a handshake. The number of steps were recorded. If the person wasn't found within 5 minutes, the task was stopped and scored as incomplete.
Time Frame: Distance to cell phone required up to 30 minutes per mode and distance to a person required up to 45 minutes per mode.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Argus II Users | Legally Blind Individuals
Number analyzed (Participants) | 4 | 5
cm
  Stationary, Normal Camera | 7 (6.6) | 4 (7.0)
  Stationary, Icon | 3 (1.8) | 4 (6.1)
  Stationary, Tone | 1 (.8) | 3 (1.5)
  Stationary, Speech | 2 (.7) | 2 (.9)
  Stationary, Normal Camera plus Tone | 3 (.5) | 1 (2.4)
  Stationary, Normal Camera plus Speech | 3. (1.6) | 1 (1.8)
  Stationary, Tone plus Icon | 1 (1.0) | 1 (.9)
  Stationary, Speech plus Icon | 2 (1.4) | 2 (1.4)
  Stationary, Tactile | 0 (0) | 0 (0)
  Mobility, Normal Camera | 52 (23.0) | 4 (4)
  Mobility, Icon | 17 (7.3) | 8 (7.5)
  Mobility, Tone | 21 (8.8) | 8 (1.6)
  Mobility, Speech | 17 (7.6) | 8 (1.7)
  Mobility, Normal Camera plus Tone | 18 (8.9) | 4 (4.0)
  Mobility, Normal Camera plus Speech | 16 (7.0) | 5 (4.5)
  Mobility, Tone plus Icon | 17 (7.8) | 6 (3.5)
  Mobility, Speech plus Icon | 17 (5.0) | 6 (3.6)

ADVERSE EVENTS:
Time Frame: 3 years
Description: Verbal reports were collected at the start of each test session, and any events occurring during the session were recorded
Arm/Group | Argus II Users | Legally Blind Individuals
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT04319809/Prot_000.pdf
  • Informed Consent Form (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/09/NCT04319809/ICF_001.pdf